CLINICAL TRIAL: NCT06769828
Title: Diagnostic Performances of Ga-68-FAPI-46 PET in CRC Patients with Rising Serum CEA During the Post-treatment Surveillance
Brief Title: Ga-68-FAPI-46 PET for CRC Recurrence Detection in Elevated CEA
Acronym: Ga-68-FAPI-46
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KF-FAPI46-001
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Recurrent
Keywords: Ga-68-FAPI-46 PET/CT; Colorectal cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga-68-FAPI-46 PET scan in colorectal cancer (Experimental): Participants in this arm will undergo a Ga-68-FAPI-46 PET scan within 2-14 days after their F-18-FDG PET scan. Ga-68-FAPI-46 will be administered via intravenous injection at a dose of 1.8-2.2 MBq per kilogram of body weight, with a maximum dose of 200 MBq. The scan will be performed 30-90 minutes after injection. This study aims to evaluate the diagnostic performance of Ga-68-FAPI-46 PET in detecting colorectal cancer recurrence in patients with elevated serum carcinoembryonic antigen (CEA), compared to F-18-FDG PET.
  Interventions: Drug: Ga-68-FAPI-46

INTERVENTIONS:
Drug: Ga-68-FAPI-46 — Ga-68-FAPI-46 PET scan in colorectal cancer
  Other Names: PET/CT

SUMMARY:
This single-center, phase II clinical trial investigates the diagnostic efficacy of Ga-68-FAPI-46 PET scans in detecting colorectal cancer (CRC) recurrence during post-treatment surveillance, particularly in patients with elevated serum carcinoembryonic antigen (CEA). The study compares the sensitivity, specificity, and accuracy of Ga-68-FAPI-46 PET with the conventional F-18-FDG PET scans, aiming to enhance recurrence detection in CRC patients who underwent curative surgery. Thirty participants will be enrolled and monitored through imaging studies and clinical follow-up.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the leading causes of cancer-related mortality, with a significant recurrence rate following curative surgery, particularly in stages II and III. Early detection of asymptomatic recurrence is critical for initiating salvage treatment. Serum CEA elevation is a marker for recurrence, necessitating advanced imaging tools for precise localization.

This study evaluates the use of Ga-68-FAPI-46, a novel imaging agent targeting fibroblast activation protein (FAP), which is overexpressed in the tumor stroma. Ga-68-FAPI-46 demonstrates higher tumor uptake and faster clearance from normal tissues compared to F-18-FDG, offering a potential diagnostic advantage. Participants will undergo both F-18-FDG PET and Ga-68-FAPI-46 PET scans, with lesion detection validated through pathology or clinical follow-up.

The trial aims to determine the diagnostic performance of Ga-68-FAPI-46 PET in terms of sensitivity, specificity, positive predictive value, and negative predictive value, using the McNemar test for statistical comparison. The study also emphasizes participant safety and data protection, adhering to Good Clinical Practice (GCP) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* The surgical intervention for colorectal cancer aims for curative resection, with the goal of achieving a disease-free status that persists for six months or more, as assessed clinically and through imaging studies.
* Elevated serum CEA levels:

Exceeding the laboratory's normal range (5 ng/ml) or, but not surpassing 13 ng/ml; using the individual's post-surgery +/- adjuvant chemotherapy or targeted therapy minimum value as a baseline, a consecutive increase of more than 10% for two times or as determined by the attending physician suggests suspicion of recurrence.

* Already performed or scheduled for FDG PET scanning examination. (5) Able to lie flat for at least 30 minutes.
* Signing the subject consent form.
* ECOG grade 0-2.
* The timing of F-18-FDG usage in this trial follows the " 2023 - Colorectal Cancer Treatment Principles" of our institution.

Exclusion Criteria:

* pregnant woman and breastfeeding women
* severe renal impairment (eGRF< 30ml/min)
* Known or suspected allergy to radiopharmaceuticals
* Simultaneously or previously diagnosed with malignant tumors other than colorectal cancer.
* Inability to undergo the necessary PET scan procedure
* Refusal or unwillingness to sign the informed consent form
* Severe medical conditions (severe disabilities, mental disorders)

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, Specificity, and Accuracy of Ga-68-FAPI-46 PET for CRC Recurrence Detection | Within 6 months of PET imaging.
  Evaluate the sensitivity, specificity, and accuracy of Ga-68-FAPI-46 PET in detecting colorectal cancer recurrence. Pathological results will be used as the reference standard where available, or clinical follow-up will be used in cases where tissue sampling is not feasible.
Comparison of Ga-68-FAPI-46 PET and FDG PET in CRC Recurrence Detection | Within 6 months of PET imaging.
  Compare the diagnostic performance of Ga-68-FAPI-46 PET and F-18-FDG PET in detecting colorectal cancer recurrence, including sensitivity, specificity, and accuracy.

SECONDARY OUTCOMES:
Clinical Impact of Ga-68-FAPI-46 PET on Management Decisions | Immediately after completion of PET imaging and report review.
  Evaluate the impact of Ga-68-FAPI-46 PET imaging on clinical decision-making through a questionnaire completed by the principal investigator before and after receiving the PET results. The questionnaire assesses changes in diagnosis, treatment planning, and patient management.

CONTACTS AND LOCATIONS:
Locations (1):
- Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Beitou, Taiwan